CLINICAL TRIAL: NCT05141253
Title: A Single-Center Exploratory Clinical Study to Evaluate the Safety and Efficacy of RD133 in Subjects With Relapsed or Refractory MSLN-Positive Solid Tumors
Brief Title: Safety and Efficacy of RD133 in Subjects With Relapsed or Refractory MSLN-Positive Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Shanghai IASO Biotechnology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-TJ-CART
Record Dates: First submitted 2021-11-09; First posted 2021-12-02 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a single center, open label, non-controlled, exploratory study. The "3+3" dose escalation design will be implemented to evaluate the safety and tolerability of RD133 in the treatment of subjects with relapsed/refractory MSLN-positive solid tumors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD133 treatment group (Experimental): Administration of RD133 Three dose groups of 1.0×10^6 CAR-T/kg, 3.0×10^6 CAR-T/kg, and 6.0×10^6 CAR-T/kg RD133 are designed in this study. 3 to 6 subjects are expected to be enrolled in each dose group according to observed DLT.
  RD133 will be intravenously infused at least 24 hours after lymphodepletion preconditioning. According to the assigned dose group, the designated dose of RD133 will be infused in a single infusion within 30 minutes on day 0.
  Interventions: Drug: RD133

INTERVENTIONS:
Drug: RD133 — The enhanced MSLN-CAR-T cell design of this study is obtained by co-infecting T cells with two lentiviral vectors. One lentiviral vector expresses CD19-CAR and tEGFR molecular safety switch, and the other lentiviral vector expresses MSLN- CAR and dnTGFβRII receptors. dnTGFβRII receptor without intracellular signal is used to resist the inhibition of T cell function by the immune microenvironment of tumor tissue. In addition, for the safety of CAR-T cell application in vivo, tEGFR is used in the CAR design as a molecular safety switch for CAR-T cells.

SUMMARY:
This study is a single-center exploratory clinical trial. It is estimated that 9-24 subjects will be enrolled. The "3+3" dose escalation design is adopted. The main purpose is to evaluate the safety of RD133 in the treatment of subjects with relapsed or refractory MSLN-positive solid tumors and explore the Recommend phase II dose of RD133 in the treatment of patients with relapsed/refractory MSLN-positive solid tumors.

DETAILED DESCRIPTION:
Leukapheresis procedure will be performed to manufacture RD133 chimeric antigen receptor (CAR) modified T cells. Bridging therapy is allowed between PBMC collection and lymphodepletion. Lymphodepletion with fludarabine and cyclophosphamide was performed for three consecutive days. After 1-day rest, subjects will receive a single dose infusion of RD133 at 1.0, 3.0, or 6.0x 10^6 CAR+ T cells/Kg. Subjects will be followed in the study for a minimum of 2 years after RD133 infusion. Long-term follow-up for lentiviral vector safety will be followed for up to 15 years after RD133 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must personally sign the written informed consent form approved by the ethics committee before the start of the study;
2. 2.≥18 years of age;
3. Have received at least 2 prior standard treatments, and achieved no response to the last-line treatment;
4. >25% Mesothelin positive rate on tumor cell membrane confirmed by prior immunohistochemistry of tumor tissue or freshly punctured tissue;
5. Expected survival ≥ 12 weeks;
6. ECOG score ≤ 2;
7. At least one measurable target lesion that meets the RECIST v1.1 standard;
8. Female or male subjects with fertility should agree to practice an effective method of contraception from the day of signing the ICF until 365 days after the infusion. Effective method of contraception is defined as: abstinence or contraceptive methods with an annual failure rate of <1% specified in the plan；
9. Before being enrolled in the group, the subject must have proper organ function and meet all of the following criteria:

9.1 The absolute value of neutrophils≥1.0×10^9/L (granulocyte colony stimulating factor (G-CSF) support is allowed, but must be without supportive treatment within 7 days before the examination); 9.2 Platelet count ≥75×10^9/L (must be without blood transfusion support [including blood component transfusion] or thrombopoietin [TPO], or other treatments for the purpose of increasing platelets within 7 days before the examination); 9.3 Hemoglobin ≥9g/dl (must be without blood transfusion support [including blood component transfusion] within 7 days before the examination); 9.4 Bilirubin value ≤1.5×upperlimit of normal (ULN) (except bile duct obstruction caused by tumor compression); 9.5 Creatinine clearance rate ≥60 ml/min; 9.6 ALT or AST≤2.5×upper limit of normal (ULN) (with liver involvement ≤5×ULN); 9.7 The results of echocardiography indicate that the cardiac ejection fraction is ≥ 50%,without obvious pericardial effusion; 9.8 Stable coagulation function: INR ≤ 1.5,APTT ≤1.2×ULN (except tumor-related anticoagulation therapy); 9.9 >91% basic blood oxygen saturation in the natural indoor air environments.

Exclusion Criteria:

1. Subject who has received any of the following prior treatments:

   1.1 Subject with acute or chronic graft-versus-host disease (GVHD) who need systemic treatment within 4 weeks before enrollment; 1.2 Subject who has received gene therapy before enrollment; 1.3 Subject who needs systematic immunosuppressive therapy (except topical drugs) to control autoimmune diseases (eg: Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, etc.), immunodeficiency or other diseases in the first 2years after enrollment; 1.4 Subject who has been injected with live vaccines within 4 weeks before enrollment; 1.5 Subject has received other interventional clinical research drugs within 12 weeks before apheresis.
2. Subject with central metastasis or complete intestinal obstruction;
3. Subject with moderate or more severe hydrothorax and ascites which are hard to control by conventional treatment and require continuous catheter drainage;
4. With an active malignant tumor in the past 5 years, unless it is a curable tumor and has been obviously cured, such as basal or squamous cell carcinoma, cervical or breast carcinoma in situ, etc.
5. Subject with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and abnormal HBV DNA test results in peripheral blood(abnormal HBV DNA test results are defined as: HBV DNA quantitative level higher than the lower limit of the detection center or higher than normal range of the detection center; or qualitative HBV DNA test positive);Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; Human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus ( CMV) DNA test positive; syphilis test RPR positive.
6. With an uncontrollable active infection (except genitourinary system infection and upper respiratory tract infection <CTCAE Grade 2).
7. Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 3), severe arrhythmia.
8. Subject with hypertension that cannot be controlled by medication.
9. The toxicity of previous treatment has not been relieved to baseline or ≤1(NCI-CTCAE v5.0, except for hair loss and laboratory abnormalities without clinical significance).
10. Major surgery within 2 weeks before enrollment, or has surgery planned during the time the subject is expected to be infused with RD133 or within12 weeks after RD133 infusion (except planned surgery under local anesthesia).
11. Subject who has a solid organ transplant.
12. Women who are pregnant or breastfeeding.
13. Subject with previous central nervous system diseases (such as cerebral aneurysm, epilepsy, stroke, Alzheimer's disease, mental illness, etc.) or mental disorders.
14. Other unstable systemic diseases judged by the investigator: including but not limited to severe liver, kidney, or metabolic diseases that require medication.
15. Known to have life-threatening allergic reactions, hypersensitivity reactions or intolerances to RD133 cell preparations or its components.
16. Subject with hemorrhage, severe thrombosis judged by the Investigator, or hereditary/acquired hemorrhage and severe thrombosis (including hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.), or are receiving thrombolytic or anticoagulant.
17. The researcher believes that other situations are not suitable for inclusion in the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2036-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Maximum of 5 years post infusion
  Type and incidence of dose-limiting toxicity (DLT) by dose group
Adverse events (AEs) and serious adverse events (SAEs) | Maximum of 5 years post infusion
  Type and incidence of adverse events (AEs) and serious adverse events (SAEs) by dose group

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values | Maximum of 5 years post infusion
  Number of Participants With Abnormal results (including laboratory tests, vital signs, physical examinations, ECG and other safety-related tests).
Objective response rate (ORR) | Maximum of 5 years post infusion
  The proportion of subjects who have achieved best response of partial response (PR) or complete response (CR) according to the RECIST V1.1evaluation criteria 3 months after RD133 cell infusion.
Duration of response (DoR) | Maximum of 5 years post infusion
  The time from the date of initial documentation of CR/PR after RD133 cell infusion to the date of progressive disease or death due to the disease studied
Time to response (TTR) | Maximum of 5 years post infusion
  The time from the date of RD133 cell infusion to the first efficacy evaluation of partial response (PR) or complete response (CR)
Disease control rate (DCR) | Maximum of 5 years post infusion
  The proportion of subjects with best efficacy assessment of complete response (CR), partial response (PR) or stable disease (SD)
Progression-free survival (PFS) | Maximum of 5 years post infusion
  The time from the date of RD133 cell infusion to the date of initial documentation of progressive disease/relapse or death from any cause.
Overall survival (OS) | Maximum of 5 years post infusion
  The time from the date of RD133 cell infusion to the date of death.
Maximum Plasma Concentration [Cmax] of RD133 in vivo | Maximum of 5 years post infusion
  Maximum Plasma Concentration [Cmax] of CAR T cell concentration in peripheral blood and tumor tissue (if any) after RD133 infusion.
Minimum Plasma Concentration [Cmin] of RD133 in vivo | Maximum of 5 years post infusion
  Minimum Plasma Concentration [Cmin] of CAR T cell concentration in peripheral blood and tumor tissue (if any) after RD133 infusion.

OTHER OUTCOMES:
TGF-β level in peripheral blood. | Maximum of 5 years post infusion
  TGF-β levels in peripheral blood after RD133 infusion.
The expression of CD3, CD4, CD8, CD68, CD163, MSLN, and PDL1 | Maximum of 5 years post infusion
  The expression of CD3, CD4, CD8, CD68, CD163, MSLN, and PDL1 in tumor tissue after RD133 cell infusion measured by Immunohistochemistry.
The positive rate of human anti-RD133 antibodies after RD133 cell infusion | Maximum of 5 years post infusion
  The proportion of patients with serum anti-RD133 antibodies after RD133 cell infusion
MSLN level in peripheral blood and in tumor tissues | Maximum of 5 years post infusion
  MSLN level in peripheral blood and in tumor tissues before and after RD133 cell infusion.
The positive rate in replication competent lentivirus (RCL). | Maximum of 5 years post infusion
  The proportion of patients with detectable replication competent lentivirus after RD133 cell infusion
T/B/NK cell ratio in peripheral blood after RD133 cell infusion. | Maximum of 5 years post infusion
  The ratio of T cell and B cell, T cell and NK cell, B cell and NK cell in peripheral blood after RD133 cell infusion.
Levels of inflammatory factors in peripheral blood after RD133 cell infusion. | Maximum of 5 years post infusion
  Levels of inflammatory factors (including but not limited to CRP, IL-6, IL-10) in peripheral blood after RD133 cell infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD. PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided